CLINICAL TRIAL: NCT05296967
Title: Efficiency of Chewing-gum to Reduce the Duration Postoperative Ileus: a Randomized Controlled Study
Brief Title: Study of the Efficience of Chewing-gum to Reduce the Duration of Postoperative Ileus
Acronym: CHEWIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Centre Hospitalier de Cholet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021_A03140_41
Record Dates: First submitted 2022-03-06; First posted 2022-03-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Ileus
MeSH Terms: interventions — Mastication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chewing gum (Experimental): POI patients are asked to chew 20 minutes x2/ day
  Interventions: Behavioral: chewing
- No chewing (No Intervention): POI patients receive no intervention

INTERVENTIONS:
Behavioral: chewing — patients are asked to chew chewing gum X 3/ day
  Arms: Chewing gum

SUMMARY:
Postoperative ileus (POI) is a serious complication after surgery. While it complicates all type of surgery, it is more frequent after abdominal surgery (especially bowel or colorectal surgery).

Many studies aim to reduce the occurence of POI without efficiency. The aim of this study is to assess the efficiency of the vagal stimulation, by the mean of chewing, to reduce the duration of POI.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing colorectal surgery or small bowel surgery
* elective or in emergency
* open surgery or laparoscopy
* diagnosis of POI
* indication of fasting or nasogastric tube placement

Exclusion Criteria:

* contra-indication of chewing
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
To assess the efficiency of chewing gum in reducing the duration of POI. POI is defined by the criteria of Vather from the postoperative day 1 up to day 30 | collected each day until the end of the POI, assessed up to day 21
  The duration of POI is the time between the first day of meeting the criteria of Vather to the day of recovery of tolerance of solid food and of exoneration of stool and/or flatus (GI-3 recovery).
  Patients will be asked to report in their diary the day of tolerance of solid food and of exoneration of stool and/or flatus (GI-3 recovery) after the diagnosis of POI

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - University Hospital aof Angers, Angers
  - CH Château Gontier, Château-Gontier
  - CH Cholet, Cholet
  - CHD Vendée, La Roche-sur-Yon
  - CH Laval, Laval
  - CHU Nantes, Nantes

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol
Time Frame: The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement.
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).